CLINICAL TRIAL: NCT01017276
Title: A Phase 3 Study in Patients With Chronic Kidney Disease (CKD) With Hyperphosphatemia on Peritoneal Dialysis
Brief Title: A Phase 3 Study in Patients With Chronic Kidney Disease and Hyperphosphatemia on Peritoneal Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1585-CL-0005
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Last update posted 2015-05-04 (Estimated); Status verified 2015-04

CONDITIONS: Chronic Kidney Disease; Renal Dialysis; Renal Insufficiency
Keywords: Hyperphosphatemia; Peritoneal dialysis; CKD; ASP1585
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Hyperphosphatemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASP group (Experimental)
  Interventions: Drug: ASP1585

INTERVENTIONS:
Drug: ASP1585 — oral
  Other Names: ILY101; AMG223

SUMMARY:
This is a multi-center, open-labeled, non-comparative study to examine the safety and efficacy of ASP1585 in chronic kidney disease and hyperphosphatemia patients on peritoneal dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients on peritoneal dialysis
* Hyperphosphatemia
* Patients on a phosphate binder or phosphate lowering drug for 28 days or longer, and that, those for whom the dose has not changed within 28 days.
* Written informed consent

Exclusion Criteria:

* Patients with gastrointestinal surgery or enterectomy
* Patients with severe cardiac diseases
* Patients with severe constipation or diarrhea
* Patients with a history or complication of malignant tumors
* Patients with uncontrolled hypertension
* Patients treated with parathyroid intervention

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Serum phosphorus level at treatment discontinuation | During the 12-week treatment period

SECONDARY OUTCOMES:
Percent of the patients meeting the target range of serum phosphorus levels | During treatment
Time-course changes in serum calcium levels | During Treatment
Changes in serum Ca x P | During Treatment
Changes in intact PTH levels | During Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Chair — Astellas Pharma Inc
Locations (3):
- Japan (3):
  - Chugoku
  - Chūbu
  - Kantou